CLINICAL TRIAL: NCT05271305
Title: Pilot Study for a National Screening for Familial Hypercholesterolemia
Acronym: EARLIE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Centre Hospitalier du Luxembourg (Other)
Collaborators: Luxembourg Institute of Health (Other Government)
Responsible Party: Principal Investigator, Carine de Beaufort, professor pediatrics, Centre Hospitalier du Luxembourg
Other Study IDs: FHC
Record Dates: First submitted 2022-02-23; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A pilot study to study the feasibility of the screening of familial hypercholesterolemia within the setting of the legal medical visits at primary school.

The pilot study shall evaluate whether this screening set-up is efficient to detect patients having familial hypercholesterolemia, detect further patients by an adjacent cascade screening of family members, to deliver treatment to these patients and to provide this screening in a cost-effective manner.

DETAILED DESCRIPTION:
Pilot study evaluating the feasibility of a screening for familial hypercholesterolemia.

Cross-sectional design. Primary outcome Percentage of screened school children with confirmed familial hypercholesterolemia Participants All children, who attend a public primary school in the city of Luxembourg and are enrolled in the cycle C2.2 (age of 7-8 years; 3rd medical visit at school), cycle C3.2 (age 9-10 years, 4th medical visit at school) and cycle 4.2 (age 11-12 years, 5th medical visit at school) will be invited to participate. Expected number of invited children is around 1600 children/year.

Recruitment will take place during the school year 2021/2022 and 2022/2023. The parents/caregivers of these children will receive written information about the screening. They will receive as well a questionnaire on the family history of premature cardiovascular events and known FHC disease.

Without informed consent, the child cannot be included in the screening program.

All children with signed informed consent will have a finger prick for a capillary blood test in the setting of their medical school exam by an external study nurse (not the school nurse) All data (pseudonymised) on each participant will be entered in the online data base for further analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Attending primary school in the city of Luxembourg and invited for the legal medical visit

Exclusion Criteria:

1. No parental informed consent

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All children, invited for their medical check through school medicine unit of the city of luxembourg, are invited to participate
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-09-04 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
familial hypercholesteromia | 2021-2024
  percentage of screened primary school children with hypercholesterolemia

SECONDARY OUTCOMES:
percentage of children screened | 2021-2024
  number screened/number invited
percentage of families screened | 2021-2024
  index case family screening

CONTACTS AND LOCATIONS:
Overall Officials: Carine de Beaufort, MPhD, Principal Investigator — CHL; Marianne Becker, MD, Principal Investigator — CHL
Locations (1):
- CHde Luxembourg, Luxembourg, Luxembourg

REFERENCES:
- [Derived] Becker M, Adamski A, Fandel F, Vaillant M, Wagner K, Droste DW, Ziade B, Hein S, Mendon P, Bocquet V, de Beaufort C. Screening for familial hypercholesterolaemia in primary school children: protocol for a cross-sectional, feasibility study in Luxembourg city (EARLIE). BMJ Open. 2022 Dec 9;12(12):e066067. doi: 10.1136/bmjopen-2022-066067. PMID 36600332